CLINICAL TRIAL: NCT01395524
Title: A Randomized, Double-Blind, Placebo-Controlled 12-Week Extension Study to Assess the Safety and Tolerability of NKTR-118 in Patients With Non-Cancer-Related Pain and Opioid-Induced Constipation (OIC)
Brief Title: A 12-week Extension of the Phase III Study (D3820C00004) to Assess the Effect and Safety of NKTR-118 in Patients With Non-cancer-related Pain and Opioid-induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3820C00007
Record Dates: First submitted 2011-06-28; First posted 2011-07-15 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Opioid-Induced Constipation (OIC)
Keywords: Non-Cancer-Related Pain; Opioid-Induced Constipation.
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NKTR-118 12.5mg (Experimental)
  Interventions: Drug: NKTR-118
- NKTR-118 25mg (Experimental)
  Interventions: Drug: NKTR-118
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-118 — 12.5 mg oral tablet once daily
  Arms: NKTR-118 12.5mg
Drug: NKTR-118 — 25 mg oral tablet once daily
  Arms: NKTR-118 25mg
Drug: Placebo — Oral tablet intake once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect and safety of NKTR-118 treatment of opioid-induced constipation in patients with non-cancer-related pain over a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the 12-week study D3820C00004 through Visit 8.
* Provision of written informed consent prior to any study-specific procedures.
* Men and women who were between the ages of >18 and <85 years at the time of the screening visit for study D3820C00004.
* Continuing to receive a stable maintenance opioid regimen consisting of a total daily dose of 30 mg to 1000 mg of oral morphine, or equianalgesic amount(s) of 1 or more other opioid therapies.
* Willingness to continue abstinence from all laxatives and other bowel regimens including prune juice and herbal products throughout this additional 12-week treatment period, and to use only bisacodyl as rescue medication if a bowel movement (BM) has not occurred within at least 72 hours of the last recorded BM.

Exclusion Criteria:

* Patients receiving opioid regimen for treatment of pain related to cancer.
* History of cancer within 5 years from the screening visit of study D3820C00004 with the exception of basal cell cancer and squamous cell skin cancer.
* Medical conditions and treatments associated with diarrhea, intermittent loose stools, or constipation.
* Other issues related to the gastrointestinal tract that could impose risk to the patient.
* Pregnancy or lactation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca
Locations (116):
- United States (90):
  - Research Site, Birmingham, Alabama
  - Research Site, Calera, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Malvern, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Garden Grove, California
  - Research Site, Laguana Hills, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Gatos, California
  - Research Site, Montebello, California
  - Research Site, National City, California
  - Research Site, Norwalk, California
  - Research Site, Paramount, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Denver, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Crystal River, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Orlando, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Venice, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Bloomington, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Reserach Site, Indianapolis, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Pikesville, Maryland
  - Research Site, Brockton, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Biloxi, Mississippi
  - Research Site, Saint Joseph, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Trenton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Beavercreek, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Medord, Oregon
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Huntingdon Valley, Pennsylvania
  - Research Site, Levittown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Yardley, Pennsylvania
  - Research Site, Cumberland, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Clarksville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Doral, Texas
  - Research Site, Houston, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Spokane, Washington
- Australia (8):
  - Research Site, Broadmeadow, New South Wales
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Port Kembla, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Greenslopes, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Fremantle, Western Australia
  - Research Site, Nedlands, Western Australia
- Germany (14):
  - Research Site, Potsdam, BR
  - Research Site, Hamburg, Hamburg
  - Research Site, Dietzenbach, Hesse
  - Research Site, Hüttenberg, Hesse
  - Research Site, Wetzlar, Hesse
  - Research Site, Celle, Lower Saxony
  - Research Site, Hanover, Lower Saxony
  - Research Site, Schwerin, Mecklenburg-Vorpommern
  - Research Site, Essen, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Leipzig, Saxony
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Berlin
  - Research Site, Dresden
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Prešov

REFERENCES:
- [Background] Webster L, Tummala R, Diva U, Lappalainen J. A 12-week extension study to assess the safety and tolerability of naloxegol in patients with noncancer pain and opioid-induced constipation. J Opioid Manag. 2016 Nov/Dec;12(6):405-419. doi: 10.5055/jom.2016.0360. PMID 28059433
- [Derived] Lawson R, King F, Marsh K, Altincatal A, Cimen A. Impact of Treatment with Naloxegol for Opioid-Induced Constipation on Patients' Health State Utility. Adv Ther. 2016 Aug;33(8):1331-46. doi: 10.1007/s12325-016-0365-y. Epub 2016 Jun 24. PMID 27342744
- See also: Clinical_Study_Report_Synopsis_D3820C00007 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1389&filename=Clinical_Study_Report_Synopsis_D3820C00007.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in the United States between 07 July 2011 and 13 September 2012.
Pre-assignment Details: Study D380C00007 is an extension study of D3820C00004. Of the patients randomized in D3820C00004, n=302 continued and enrolled into D380C00007. The study duration was up to 14 weeks, consisting of a 12 week treatment period and a follow-up visit 2 weeks after the last dose of study drug.
Groups:
- NKTR-118 12.5 mg: NKTR-118 12.5 mg QD, oral treatment
- NKTR-118 25 mg: NKTR-118 25 mg QD, oral treatment
- Placebo: Placebo QD, oral treatment
Period: Overall Study
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Started | 97 | 99 | 106
Completed | 79 | 83 | 89
Not Completed | 18 | 16 | 17
Not completed — Non-compliance with study schedule | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Study-Specific Withdrawal Criteria | 1 | 2 | 0
Not completed — Severe noncompliance with protocol | 1 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Eligibility Criteria Not Fulfilled | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 8
Not completed — Did not receive treatment | 1 | 1 | 3
Not completed — Subject had spinal surgery | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 6 patients (1 patient in the NKTR-118 25 mg group, 2 patients in the NKTR-118 12.5 mg group, 3 patients in the placebo group) had been previously randomized within the NKTR-118 program at a different study center and were excluded from the ITT and Safety analysis sets. Baseline characteristics are summarized using the ITT analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo | Total
Number analyzed (Participants) | 95 | 98 | 103 | 296
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (9.51) | 52.6 (10.19) | 52.6 (10.00) | 52.3 (9.89)
Gender [Count of Participants; unit: Participants]
  Female | 62 | 57 | 61 | 180
  Male | 33 | 41 | 42 | 116
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 71 | 74 | 76 | 221
  Black or African American | 24 | 22 | 23 | 69
  Asian | 0 | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Other | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Patients Experiencing at Least One Adverse Event (AE)
Description: The incidence of patients experiencing at least one AE during the randomized treatment and follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period (Week 14)
Population: The Safety analysis set included all patients who participated in Study D3820C00004 and received at least 1 dose of study drug in Study D3820C00007, with the exception of patients who were found to have randomized multiple times within the program at different centers.
Measure: Number; unit: Participants
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 94 | 97 | 100
Participants | 32 | 40 | 33

2. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Symptoms Questionnaire (PAC-SYM)
Description: The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe) in the 2 weeks (14 days) prior to assessment. Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range of the domain or total score is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (prior to treatment) to last on-treatment assessment (up to Week 12)
Population: The modified intent-to-treat(ITT) analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers. The N denotes the number of patients with a baseline and last on-treatment value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 84 | 90 | 97
units on a scale
  Total score | -0.9 (0.71) | -0.9 (0.85) | -0.8 (0.84)
  Abdominal symptoms subscore | -0.8 (0.85) | -0.7 (0.97) | -0.7 (0.82)
  Rectal symptoms subscore | -0.7 (0.84) | -0.7 (0.84) | -0.6 (0.90)
  Stool symptoms subscore | -1.2 (0.90) | -1.1 (1.04) | -0.9 (1.04)

3. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Quality of Life (PAC-QOL)
Description: The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being in the 2 weeks (14 days) prior to assessment. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) Worries and concerns (11 items), 2) Physical discomfort (4 items), 3) Psychosocial discomfort (8 items), and 4) Satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range of the domain or total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (prior to treatment) to last on-treatment assessment (up to Week 12)
Population: The modified intent-to-treat (ITT) analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers.The N denotes the number of patients with a baseline and last on-treatment value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 84 | 89 | 96
units on a scale
  Total score | -1.0 (0.89) | -0.9 (0.82) | -0.8 (0.74)
  Physical discomfort | -1.0 (0.97) | -1.1 (0.97) | -1.0 (0.96)
  Psychosocial discomfort | -0.8 (0.97) | -0.7 (0.86) | -0.6 (0.81)
  Worries/concerns | -1.0 (1.09) | -0.9 (0.91) | -0.7 (0.86)
  Satisfaction | -1.2 (1.14) | -1.3 (1.22) | -1.1 (1.21)

4. Primary Outcome: Incidence of Patients Experiencing AEs That Resulted in Discontinuation of Investigational Product (IP)
Description: The incidence of patients experiencing AEs that resulted in discontinuation of IP during the randomized treatment or follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period (Week 14)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 94 | 97 | 100
Participants | 4 | 4 | 3

5. Primary Outcome: Incidence of Patients Experiencing Severe Adverse Events (SAEs)
Description: The incidence of patients experiencing SAEs during the randomized treatment and follow-up periods was calculated.
Time Frame: Baseline (Week 0) to end of the follow-up period (Week 14)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 94 | 97 | 100
Participants | 6 | 6 | 5

ADVERSE EVENTS:
Description: Safety population, i.e. patients who received at least one dose of study medication, was used as the At Risk population
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/94 | 6/97 | 5/100
Other Adverse Events (participants affected / at risk) | 15/94 | 27/97 | 11/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=94) | NKTR-118 25 mg (N=97) | Placebo (N=100)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 (1) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILU RE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=94) | NKTR-118 25 mg (N=97) | Placebo (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
LOCAL SWELLING (General disorders) | 0 (0) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
SINUSITIS (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
BLOOD TESTOSTERONE DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days